CLINICAL TRIAL: NCT06791941
Title: Study of the Contribution of Mutant p53/YAP Proteins to Therapy Resistance in Recurrent Head and Neck Cancer
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS105/IRE/24
Record Dates: First submitted 2025-01-16; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Tumors
Keywords: head and neck tumors; TP53; organoids
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Extraction of RNA and DNA from fresh tissue samples, and paraffin-embedded tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Culture of organoids — Culture of organoids prepared from both the primary tumor and the respective relapse, using the material from the prospective part of the study, the response to treatment will be carried out by macroscopic analysis, evaluating the size and number of organoids before and after treatment,

SUMMARY:
Multicenter, non-interventional, retrospective/prospective study of a biological nature, on patients affected by head and neck tumors, for which the collection and use of tissue samples is planned for the study of the mutational profile, the transcriptional profile and the proteomic profile.

DETAILED DESCRIPTION:
The study aims to characterize molecular networks governed by the mutated protein p53 with a relevant role in the development of local recurrence in head and neck tumors HNSCC, in order to identify the main actors involved in resistance to current therapy and try to develop new more effective therapeutic strategies for head and neck tumors.

Furthermore, the existence of a significant relationship between the time of onset of recurrence and the deregulation of the identified molecular networks will be studied.

This study will therefore allow to:

1. Identify networks associated with the presence of mutation in the TP53 gene relevant in the development of relapse, comparing the tissues of the primary tumor to the respective tissue of the relapse of patients affected by head and neck cancer, by:

   1. expression profiles of coding and non-coding RNAs (retrospective cohort)
   2. mutational profile by NGS (retrospective cohort)
   3. Single cell RNA-sequencing (SC-RNAseq) on samples belonging to the prospective cohort
2. Characterize the molecular mechanisms underlying TP53-dependent networks with a key role in resistance to therapy, using resistance cell systems and in organoid cultures derived from head and neck tumors HNSCC (PDO) (prospective cohort).
3. Identify the best treatment combinations able to target the networks identified as associated with resistance (prospective cohort).
4. To evaluate the response of treatments in vivo using a syngeneic model of head and neck tumors HNSCC (MOC model).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patients with squamous cell tumors of the oral cavity, pharynx or larynx
* Surgical patients with primary HNSCC tumors, who have not had previous tumors in other sites or adjuvant treatments prior to surgery.
* Availability of adequate material (tissue) for the planned analyses
* Availability of follow-up data for at least one year (retrospective part)
* Written informed consent (prospective part and/or, for the retrospective part, traceable patients and/or patients in follow-up and/or if necessary for the legal nature/institutional purposes of the participating centers).

Exclusion Criteria:

* Presence of distant metastases at the time of diagnosis
* Previous head and neck cancer
* Second cancer undergoing treatment or follow-up for less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck tumors
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2029-03-07 (Estimated); Study Completion 2029-03-07 (Estimated)

PRIMARY OUTCOMES:
Organoids cultures | 60 months
  Fresh tissue samples collected from surgery at the reference centers will be selected by the pathologist, and stored at 4°C in special media at the reference laboratories. These samples will be evaluated by means of viabilityassays with ATPlite, the ability to form colonies and apoptosis assays (by FACS). For organoids, the response to treatment will be performed by macroscopic analysis, evaluating the size and number of organoids before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Blandino, Doctor, Principal Investigator — IRCCS National Cancer Institute
Locations (1):
- IRCCS National Cancer institute, Roma, Rome, Italy